CLINICAL TRIAL: NCT03578081
Title: Olanzapine With or Without Fosaprepitant for the Prevention of Chemotherapy Induced Nausea and Vomiting (CINV)in Patients Receiving Highly Emetogenic Chemotherapy (HEC): A Phase III Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Olanzapine With or Without Fosaprepitant Dimeglumine in Preventing Chemotherapy Induced Nausea and Vomiting in Cancer Patients Receiving Highly Emetogenic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A221602; NCI-2017-02410 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-05 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Palonosetron; Ondansetron; Dexamethasone; fosaprepitant; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (fosaprepitant dimeglumine, olanzapine) (Experimental): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, fosaprepitant dimeglumine IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Palonosetron Hydrochloride; Drug: Ondansetron Hydrochloride; Drug: Dexamethasone; Drug: Fosaprepitant Dimeglumine; Drug: Olanzapine
- Arm II (placebo, olanzapine) (Active Comparator): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, placebo IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment (with no placebo) may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Palonosetron Hydrochloride; Drug: Ondansetron Hydrochloride; Drug: Dexamethasone; Drug: Olanzapine; Other: Placebo

INTERVENTIONS:
Drug: Palonosetron Hydrochloride — Given IV
Drug: Ondansetron Hydrochloride — Given IV or PO
Drug: Dexamethasone — Given PO
Drug: Fosaprepitant Dimeglumine — Given IV
  Arms: Arm I (fosaprepitant dimeglumine, olanzapine)
Drug: Olanzapine — Given PO
Other: Placebo — Given IV
  Arms: Arm II (placebo, olanzapine)

SUMMARY:
This randomized phase III trial studies how well olanzapine with or without fosaprepitant work in preventing chemotherapy induced nausea and vomiting in cancer patients receiving chemotherapy that causes vomiting. Olanzapine and fosaprepitant dimeglumine may help control nausea and vomiting in patients during chemotherapy. Olanzapine is usually given in combination with other drugs, including fosaprepitant dimeglumine. It is not yet known if olanzapine when given with other drugs, is still effective without using fosaprepitant dimeglumine for controlling nausea and vomiting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare between the two study arms the proportion of patients with no nausea for the overall (0-120 hours post-chemotherapy), acute (0-24 hours post-chemotherapy), and delayed periods (24-120 hours post-chemotherapy) for patients receiving highly emetogenic chemotherapy (HEC).

SECONDARY OBJECTIVES:

I. To compare between the two study arms the complete response (CR) rates (no emetic episodes and no use of rescue medication) in the acute, delayed, and overall periods.

II. To compare between the two study arms, the incidences of potential toxicities that have been ascribed to olanzapine.

III. To perform an economic evaluation of olanzapine and fosaprepitant dimeglumine (fosaprepitant) versus (vs.) olanzapine in patients receiving HEC (noting that all patients will also receive dexamethasone and a 5HT3 receptor antagonist).

IV. To explore the efficacy of olanzapine in chemotherapy cycles two to four, for patients who elect to continue on the same antiemetic regimen received in cycle one, in chemotherapy cycles two to four (continuation phase), by documenting nausea and complete response.

V. To explore the safety of olanzapine in chemotherapy cycles two to four, for patients who elect to continue on the same antiemetic regimen received in cycle one, in chemotherapy cycles two to four (continuation phase), by recording any adverse events or drug related toxicities.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive palonosetron hydrochloride intravenously (IV) over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or orally (PO) on day 1, dexamethasone PO on days 1-4, fosaprepitant dimeglumine IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, placebo IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment (with no placebo) may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant disease of any stage; (stage I through stage IV)
* No prior history of chemotherapy for any malignancy
* Scheduled to receive intravenous HEC (highly emetogenic chemotherapy) (either cisplatin-containing regimen or doxorubicin and cyclophosphamide [AC]); cisplatin, given on a single day, at a dose of >= 70 mg/m^2, with or without other chemotherapy agent(s) OR doxorubicin (60 mg/m^2) plus cyclophosphamide (600 mg/m^2)
* No nausea or vomiting =< 24 hours prior to registration
* Negative pregnancy test (serum or urine) done =< 7 days prior to registration, for women of childbearing potential only

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* No known diagnosis of dementia; patients with stable treated brain metastases are eligible to participate
* No known history of central nervous system (CNS) disease (e.g. seizure disorder)
* No treatment with another antipsychotic agent such as olanzapine, risperidone, quetiapine, clozapine, phenothiazine or butyrophenone =< 30 days prior to registration
* No chronic phenothiazine administration as an antipsychotic agent (patients may receive prochlorperazine and other phenothiazines as rescue anti-emetic therapy but not within 24 hours prior to registration)
* No use of amifostine within 7 days prior to registration
* No radiotherapy within 7 days prior to registration or planned for one week after the current dose of chemotherapy
* No use of quinolone antibiotic therapy within 7 days prior to registration
* No chronic alcoholism (as determined by the investigator)
* No known hypersensitivity to olanzapine
* No known uncontrolled cardiac arrhythmia, no known uncontrolled congestive heart failure, or no acute myocardial infarction within the previous six months
* No history of uncontrolled diabetes mellitus, i.e., no diabetic ketoacidosis; within 6 months prior to registration; patients are eligible if they have controlled diabetes on diet, oral agents, and/or insulin
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Patients must be able to read and comprehend English; local translation, including verbal translation of patient-reported outcomes (PROs) is not permitted
* Serum creatinine =< 2.0 mg/dL =< 120 days prior to registration
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN) =< 120 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolph Navari, MD, PhD, FACP, Study Chair — University of Alabama at Birmingham
Locations (566):
- United States (565):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - MercyOne Waterloo Medical Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Saint Claire Regional Medical Center, Morehead, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Ochsner LSU Health Saint Mary's Medical Center, Shreveport, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Cancer Partners of Nebraska - Pine Lake, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center - 68th Street Place, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - CarolinaEast Oncology and Hematology Associates, New Bern, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- FHP Health Center-Guam, Tamuning, Guam

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data Set
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Navari RM, Le-Rademacher J, Smieliauskas F, Ruddy KJ, James Saphner T, Liu H, Harlos E, Onitilo AA, Giridhar K, Paul Singh P, Reddy PS, Chow S, Kruter F, Raptis G, Loprinzi CL. Olanzapine With or Without Fosaprepitant for Preventing Chemotherapy Induced Nausea and Vomiting in Patients Receiving Highly Emetogenic Chemotherapy: A Phase III Randomized, Double-Blind, Placebo-Controlled Trial (ALLIANCE A221602). Oncologist. 2023 Aug 3;28(8):722-729. doi: 10.1093/oncolo/oyad140. PMID 37284847
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Fosaprepitant Dimeglumine, Olanzapine): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, fosaprepitant dimeglumine IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.>>
  >> Palonosetron Hydrochloride: Given IV>>
  >> Ondansetron Hydrochloride: Given IV or PO>>
  >> Dexamethasone: Given PO>>
  >> Fosaprepitant Dimeglumine: Given IV>>
  >> Olanzapine: Given PO
- Arm II (Placebo, Olanzapine): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, placebo IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment (with no placebo) may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.>>
  >> Palonosetron Hydrochloride: Given IV>>
  >> Ondansetron Hydrochloride: Given IV or PO>>
  >> Dexamethasone: Given PO>>
  >> Olanzapine: Given PO>>
  >> Placebo: Given IV
Period: Overall Study
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine)
Started | 346 | 344
Completed | 326 | 320
Not Completed | 20 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine) | Total
Number analyzed (Participants) | 346 | 344 | 690
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.10) | 56.1 (11.58) | 56.3 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289 | 289 | 578
  Male | 57 | 55 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 331 | 325 | 656
  Unknown or Not Reported | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 4 | 12 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 36 | 40 | 76
  White | 292 | 278 | 570
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 12 | 11 | 23
ECOG Performance Score [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction.> ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.> ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.> ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 276 | 281 | 557
    1 | 67 | 59 | 126
    2 | 3 | 4 | 7
Chemotherapy Regimen [Count of Participants; unit: Participants]
  Anthracycline and cyclophosphamide (AC) | 267 | 266 | 533
  Cisplatin-containing regimen | 79 | 78 | 157
5-HT Receptor Antagonist [Count of Participants; unit: Participants]
  Ondansetron | 90 | 90 | 180
  Palonosetron | 256 | 254 | 510

OUTCOME MEASURES:

1. Primary Outcome: No Nausea Rate Defined as a Response of 0 in the Nausea Item of Nausea and Vomiting Daily Diary/Questionnaire in the Overall (0-120 Hours), Acute (0-24 Hours), and Delayed (24-120 Hours) Periods
Description: The specific measure will be based on the proportion of patients with a value of 0, as measured by the single nausea item (scale 0-10, 0 is no symptoms, 10 is worst symptoms) of the Questionnaire. A modified intent-to-treat principle will be applied for statistical analysis of efficacy in evaluable patients. The proportions of patients with no nausea during the overall, the acute, and the delayed period will be summarized by treatment arm. They will be tested in a sequential manner, using a Simes gatekeeping procedure to maintain the overall significance level at the specified by the Lan-DeMets family of alpha spending function. The difference in no nausea proportions between arms will be estimated along with a one-sided 95% confidence interval. The tests and the confidence intervals will be constructed using normal approximation of the binomial distribution adjusted for the non-inferiority margin.
Time Frame: Up to 120 hours
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Fosaprepitant Dimeglumine, Olanzapine): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, fosaprepitant dimeglumine IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Palonosetron Hydrochloride: Given IV>
  >>
  >
  >> Ondansetron Hydrochloride: Given IV or PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Fosaprepitant Dimeglumine: Given IV>
  >>
  >
  >> Olanzapine: Given PO
- Arm II (Placebo, Olanzapine): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, placebo IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment (with no placebo) may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Palonosetron Hydrochloride: Given IV>
  >>
  >
  >> Ondansetron Hydrochloride: Given IV or PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Olanzapine: Given PO>
  >>
  >
  >> Placebo: Given IV
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine)
Number analyzed (Participants) | 326 | 320
Participants
  Overall No Nausea | 123 | 97
  Overall Any Nausea | 203 | 223
  Acute No Nausea | 202 | 201
  Acute Any Nausea | 124 | 119
  Delayed No Nausea | 140 | 114
  Delayed Any Nausea | 186 | 206

2. Secondary Outcome: Complete Response (CR) (no Emetic Episodes and no Use of Rescue Medication) During the Acute, Delayed and the Overall Periods as Measured by the Nausea and Vomiting Daily Diary/Questionnaire
Description: The specific measure will be based on the proportion of patients who answered "None" to both questions concerning Vomiting episode(None, Once, Twice, More than twice) and number of extra nausea/vomiting pills taken (None, One, Two, More than two) in the Nausea and Vomiting Daily Diary/Questionnaire. The CR rate for the overall, the acute, and the delayed period will be summarized by treatment arm and will be compared using a Chi-squared test. The difference in CR rates between arms will be estimated along with a 95% confidence interval.
Time Frame: Up to 120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine)
Number analyzed (Participants) | 326 | 320
Participants
  Complete Response - >> Overall | 179 | 151
  Complete Response - >> Acute | 256 | 247
  Complete Response ->> Delayed | 193 | 166

3. Secondary Outcome: Potential Toxicities as Ascribed to Olanzapine as Measured by the Nausea and Vomiting Daily Diary/Questionnaire
Description: Potential toxicities includes nausea, undesired sedation, and undesired appetite, measured by three individual items ( nausea, undesired sedation, undesired appetite) of the Nausea and Vomiting Daily Dairy/Questionnaire(scale 0-10, 0 is no symptoms, 10 is worst symptoms). Incidences of toxicities will be summarized by type and by treatment arm. Incidences of toxicities will be compared between arms using a Chi-squared test or the Fisher's exact test as appropriate. In addition, undesired sedation and appetite increase as collected in the Nausea and Vomiting Daily Diary/Questionnaire will be analyzed by repeated measures analyses including descriptive statistics, graphical approaches, and growth curve models to account for the factor of day and time trend.
Time Frame: Up to 120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine)
Number analyzed (Participants) | 326 | 320
Participants
  Overall No Appetite Increase | 140 | 136
  Overall Any Appetite Increase | 186 | 184
  Acute No Appetite Increase | 235 | 236
  Acute Any Appetite Increase | 91 | 84
  Delayed No Appetite Increase | 147 | 143
  Delayed Any Appetite Increase | 179 | 177

4. Secondary Outcome: Average Nausea Scores (0-10) Repeatedly Measured by the Nausea and Vomiting Daily Diary/Questionnaire
Description: The specific measure will be based on the by the single nausea item (scale 0-10, 0 is no symptoms, 10 is worst symptoms) of the Nausea and Vomiting Daily Diary/Questionnaire. Nausea scores (0-10) repeatedly measured by the Nausea and Vomiting Daily Diary/Questionnaire will be analyzed using the repeated measures analyses and growth curve models as described above for undesired sedation and increase in appetite.
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine)
Number analyzed (Participants) | 326 | 320
score on a scale | 0.8211364 (1.6289005) | 0.9177778 (1.7821806)

5. Secondary Outcome: Total Frequency of Rescue Medication as Measured by the Nausea and Vomiting Daily Diary/Questionnaire
Description: The specific measure will be based on the single item : number of extra nausea/vomiting pills taken (None, One , Twice, More than twice) of the Nausea and Vomiting Daily Diary/Questionnaire.
Time Frame: Over 5 Days per each of the 4 cycles
Measure: Number; unit: episodes
Groups:
- Arm I (Fosaprepitant Dimeglumine, Olanzapine): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, fosaprepitant dimeglumine IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > Palonosetron Hydrochloride: Given IV
  >
  >
  >
  >
  >
  > Ondansetron Hydrochloride: Given IV or PO
  >
  >
  >
  >
  >
  > Dexamethasone: Given PO
  >
  >
  >
  >
  >
  > Fosaprepitant Dimeglumine: Given IV
  >
  >
  >
  >
  >
  > Olanzapine: Given PO
- Arm II (Placebo, Olanzapine): Patients receive palonosetron hydrochloride IV over 30 seconds or ondansetron hydrochloride IV over 2-5 minutes or PO on day 1, dexamethasone PO on days 1-4, placebo IV over 20-30 minutes on day 1, and olanzapine PO on days 1-4. Treatment (with no placebo) may repeat every 4 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > Palonosetron Hydrochloride: Given IV
  >
  >
  >
  >
  >
  > Ondansetron Hydrochloride: Given IV or PO
  >
  >
  >
  >
  >
  > Dexamethasone: Given PO
  >
  >
  >
  >
  >
  > Olanzapine: Given PO
  >
  >
  >
  >
  >
  > Placebo: Given IV
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine)
Number analyzed (Participants) | 326 | 320
episodes
  Zero | 3614 | 3541
  One | 350 | 405
  Two | 170 | 162
  More than two | 56 | 74

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Arm I (Fosaprepitant Dimeglumine, Olanzapine) | Arm II (Placebo, Olanzapine)
All-Cause Mortality (participants affected / at risk) | 1/286 | 2/291
Serious Adverse Events (participants affected / at risk) | 51/286 | 60/291
Other Adverse Events (participants affected / at risk) | 252/286 | 248/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Fosaprepitant Dimeglumine, Olanzapine) (N=286) | Arm II (Placebo, Olanzapine) (N=291)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 9 (9) | 10 (10)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 5 (5) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Fosaprepitant Dimeglumine, Olanzapine) (N=286) | Arm II (Placebo, Olanzapine) (N=291)
Anemia (Blood and lymphatic system disorders) | 13 (13) | 18 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 19 (19) | 22 (22)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 3 (3) | 5 (5)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Thrush (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 20 (20) | 17 (17)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 20 (20) | 19 (19)
Platelet count decreased (Investigations) | 3 (3) | 7 (7)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 11 (11) | 17 (17)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 11 (11) | 15 (15)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14) | 20 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03578081/Prot_SAP_ICF_001.pdf